CLINICAL TRIAL: NCT02514122
Title: Subcutaneous Ketamine for Postoperative Pain Relief in Rwanda: a Randomized Control Trial
Brief Title: Subcutaneous Ketamine for Postoperative Pain Relief in Rwanda
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: National University, Rwanda (Other)
Responsible Party: Principal Investigator, William McKay, MD FRCPC, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio# 14-193
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Post Operative Pain; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Participants will receive subcutaneous ketamine (1mg/kg) administered immediately after surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections at a dose of 1mg/kg.
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): Participants will receive subcutaneous saline (0.02cc/kg) administered immediately after surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — Patients will receive a subcutaneous injection of ketamine (at a dose of 1mg/kg) immediately following surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections.
  Arms: Ketamine
Drug: Saline — Patients will receive a subcutaneous injection of saline (at a dose of 0.02cc/kg) immediately following surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections.
  Arms: Saline

SUMMARY:
A randomized double blind control trial to investigate the safety and efficacy of subcutaneous ketamine for control of post operative pain in low resource settings.

DETAILED DESCRIPTION:
A randomized double blind control trial. All patients undergoing upper abdominal, thoracic, gynecologic or orthopaedic surgeries at the Centre Hospitalier Universitaire de Kigali, Kigali, Rwanda will be invited to participate. Enrolled patients will receive subcutaneous ketamine (or placebo) administered immediately after surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections at a dose of 1mg/kg. The primary outcome will be a reduction in mean Pain Scores using parametric statistical analysis to discriminate significance. Pain will be measured using an 11-point numerical rating scale. Secondary outcomes will be the presence of significant side effects. This trial is a partnership between the University of Saskatchewan and the National University of Rwanda with ethics approval from each institutions ethics board.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing upper abdominal, thoracic, gynecologic or orthopaedic surgeries during a one month period with expected post operative hospital admission

Exclusion Criteria:

* Allergy to Ketamine
* History of narcotic abuse or dependence
* Those patients for which decreased cognitive function is a barrier to accurate data collection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Mckay, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Derived] Sacevich C, Semakuba B, McKay WP, Thakore S, Twagirumugabe T, Nyiligira J. Subcutaneous ketamine for postoperative pain relief in Rwanda: a randomized clinical trial. Can J Anaesth. 2018 Feb;65(2):170-177. doi: 10.1007/s12630-017-1009-7. Epub 2017 Nov 13. PMID 29134517

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Saline
Started | 32 | 29
Completed | 30 (one participant dropped out for religious reasons; one for needle phobia) | 29
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Saline | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.6) | 35.3 (10.8) | 38.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 11 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Rwanda | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain as Measured on a 11-point Numerical Rating Scale
Description: Pain will be measured using an 11-point numerical rating scale from 0 (no pain) to 10 (worst pain imaginable) units on a scale.
Time Frame: The average of twice daily pain scores, from end of surgery until 60 hours postoperative.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 30 | 29
units on a scale | 3.5 (1.4) | 4.9 (1.6)
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority; p = 0.009, t-test, 2 sided — The p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.29 to 1.9] — Score was lower in the Ketamine group

2. Secondary Outcome: Hallucination
Description: Presence (or not) of hallucinations.
Time Frame: From end of surgery until 60 hours postoperative.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 30 | 29
Participants
  hallucinations | 11 | 0
  no hallucination | 19 | 29
Statistical Analysis 1: Comparison: Ketamine vs Saline; Test type: Superiority; p < 0.001, Fisher Exact; Risk Difference (RD) = .37, 95% CI 2-sided [.18 to .54]

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- Ketamine: Participants will receive subcutaneous ketamine (1mg/kg) administered immediately after surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections at a dose of 1mg/kg.
  Ketamine: Patients will receive a subcutaneous injection of ketamine (at a dose of 1mg/kg) immediately following surgery, the evening after surgery, and every 12 hours thereafter for a total of 5 injections.
  Ketamine participants had more hallucinations than saline group.
Arm/Group | Ketamine | Saline
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 11/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=30) | Saline (N=30)
hallucination (Psychiatric disorders) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No